CLINICAL TRIAL: NCT06750705
Title: The Effectiveness of PechaKucha as a Reinforcement Tool in Teaching Vital Signs Skills to Nursing Students: A Randomized Controlled Trial
Brief Title: PechaKucha as a Reinforcement Tool for Teaching Vital Signs Skills in Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Nevin Doğan, DR, Siirt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 121927
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Vital Signs; Nursing Students; Teaching Method; PechaKucha Method; Skill Performance
Keywords: PechaKucha Method; Nursing Students; vital signs

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PechaKucha presentation (Experimental): This arm of the study will involve nursing students receiving reinforcement training using the PechaKucha presentation method.
  Interventions: Other: PechaKucha
- PowerPoint presentation (Active Comparator): This arm of the study will involve nursing students receiving reinforcement training using a traditional PowerPoint presentation.
  Interventions: Other: PowerPoint

INTERVENTIONS:
Other: PechaKucha — The PechaKucha format consists of 20 slides, each displayed for 20 seconds, focusing on vital signs measurement skills. The method emphasizes a fast-paced, engaging, and visual learning experience designed to enhance retention and improve students' practical knowledge and skills in measuring vital signs.
  Arms: PechaKucha presentation
Other: PowerPoint — The PowerPoint presentation will cover the same vital signs measurement content but in a more conventional, linear format. The intervention will aim to reinforce students' understanding of vital signs through text and images, with a slower pace compared to the PechaKucha method.
  Arms: PowerPoint presentation

SUMMARY:
This study aims to evaluate the effectiveness of the PechaKucha presentation method as a reinforcement tool in teaching vital signs skills to first-year nursing students. A total of 100 nursing students will participate and be divided into two groups of 50 students each. Before the intervention, all participants will complete a pre-test to assess their baseline knowledge related to vital signs. Based on the pre-test results, students will be randomized into either the experimental group or the control group.

The experimental group will receive reinforcement training using the innovative PechaKucha presentation method, while the control group will receive reinforcement through a traditional PowerPoint presentation. After the reinforcement sessions, both groups will be evaluated on their vital signs skills through a practical application exam.

Additionally, participants will complete a post-test to assess their knowledge after the intervention. Feedback and satisfaction with the training methods will also be gathered to understand their perspectives on the learning experience

DETAILED DESCRIPTION:
This study investigates the effectiveness of the PechaKucha presentation method as a reinforcement tool in teaching vital signs skills to first-year nursing students. Vital signs, including body temperature, pulse, respiration, and blood pressure, are critical indicators of a patient's overall health and play a fundamental role in early detection of health issues. Accurate measurement and interpretation of vital signs are essential for ensuring high-quality patient care and safety. Therefore, equipping nursing students with the necessary skills and confidence to perform these tasks is vital for their professional readiness in both routine and emergency healthcare scenarios.

Nursing education is a critical process aimed at developing students' knowledge, skills, and attitudes to ensure they can provide competent and high-quality healthcare services. However, traditional teaching methods often have limitations in helping students retain theoretical knowledge and translate it into practical skills. To address these limitations, innovative reinforcement methods such as PechaKucha are increasingly being incorporated into nursing education.

The PechaKucha method involves short, visually engaging presentations structured into 20 slides, each lasting 20 seconds. This rapid and interactive format has been shown to enhance students' focus, maintain their attention, and improve knowledge retention. In this study, the PechaKucha method will be compared to the traditional PowerPoint presentation approach to assess its impact on students' knowledge, skills, and satisfaction levels.

A randomized controlled trial design will be employed, involving 100 first-year nursing students divided into two groups of 50 each. Before the intervention, all participants will complete a pre-test to evaluate their baseline knowledge related to vital signs. Based on pre-test results, students will be randomized into two groups:

The experimental group, which will receive reinforcement training using the PechaKucha presentation method.

The control group, which will receive reinforcement training through a traditional PowerPoint presentation.

Following the reinforcement sessions, students' practical skills in measuring and interpreting vital signs will be evaluated through an application exam. Post-test forms will also be administered to assess their knowledge after the intervention. Feedback and satisfaction surveys will be collected to gain insights into the students' experiences with both teaching methods.

This study aims to identify whether the PechaKucha method is a more effective reinforcement tool compared to traditional methods in enhancing nursing students' learning outcomes. The findings are expected to contribute valuable insights into the use of innovative teaching methods in nursing education, with potential implications for improving the quality of training programs and ultimately ensuring better patient care outcomes.

ELIGIBILITY:
Inclusion Criteria:

* First-year nursing students currently enrolled in the nursing program.
* Students who provide informed consent to participate in the study.

Exclusion Criteria:

* Foreign nationals.
* Students repeating the course (taking the course as a retake).
* Students who have graduated from a high school or associate degree program related to healthcare.
* Students who are unable to attend the scheduled intervention sessions.
* Students with physical or cognitive impairments that would affect their ability to participate in the skills assessment or intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Vital Signs Knowledge Test | 2 days before the training
  The Vital Signs Knowledge Test is a 16-item multiple-choice questionnaire developed by the researchers to evaluate nursing students' theoretical knowledge of vital signs. The test covers essential topics such as body temperature, pulse, respiration, and blood pressure measurement procedures. Each item provides five response options, with one correct answer per question. The test is scored on a 100-point scale, with scores ranging from a minimum of 0 to a maximum of 100, where higher scores indicate a greater level of knowledge. The total score reflects the students' understanding of vital signs concepts. The test was reviewed by five experts to ensure its content validity and accuracy. It will be administered before and after the intervention to assess the students' knowledge retention and compare the effectiveness of different teaching methods (PechaKucha vs. PowerPoint) in reinforcing the learning of vital signs
Vital Signs Skills Checklist | within 1 week post-intervention assessment
  It assesses students' ability to accurately measure body temperature, pulse, respiration, and blood pressure. Each step of the procedure is scored based on its accuracy: "correctly performed," "partially correct," or "not performed." The total score will be calculated out of 100 points, with scores ranging from a minimum of 0 to a maximum of 100, where higher scores indicate a greater level of competence in vital signs measurement. The checklist has been reviewed by experts to ensure its validity and accuracy in assessing the students' competence in performing vital signs measurements
Student Feedback Form | immediately post-intervention assessment
  The Student Feedback Form will gather qualitative data on students' perceptions of the reinforcement methods. It includes two open-ended questions:
  What aspects of the reinforcement method did you like? How could the reinforcement method be improved? These questions aim to capture students' feedback on the effectiveness and potential improvements of the PechaKucha and PowerPoint methods in teaching vital signs.
Satisfaction Survey | immediately post-intervention assessment
  The Satisfaction Survey will use a visual analog scale (VAS) for students to rate their satisfaction with the reinforcement methods. Students will be asked to provide a score between 0 and 10, where 0 represents "not satisfied at all" and 10 represents "extremely satisfied." The survey is scored on a scale from a minimum of 0 to a maximum of 10, with higher scores indicating greater levels of satisfaction. This survey will assess students' overall satisfaction with the PechaKucha and PowerPoint methods in terms of their learning experience and perceived effectiveness in reinforcing vital signs skills.
Vital Signs Knowledge Test | within 1 week post-intervention assessment
  The Vital Signs Knowledge Test is a 16-item multiple-choice questionnaire developed by the researchers to evaluate nursing students' theoretical knowledge of vital signs. The test covers essential topics such as body temperature, pulse, respiration, and blood pressure measurement procedures. Each item provides five response options, with one correct answer per question. The test is scored on a 100-point scale, with scores ranging from a minimum of 0 to a maximum of 100, where higher scores indicate a greater level of knowledge. The total score reflects the students' understanding of vital signs concepts. The test was reviewed by five experts to ensure its content validity and accuracy. It will be administered before and after the intervention to assess the students' knowledge retention and compare the effectiveness of different teaching methods (PechaKucha vs. PowerPoint) in reinforcing the learning of vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Nevin Doğan, Principal Investigator — Siirt University
Locations (1):
- Siirt University, Siirt, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dogan N, Aksoy M. The effectiveness of PechaKucha as a reinforcement tool in teaching vital signs skills to nursing students: A randomized controlled trial. Nurse Educ Today. 2026 Jan;156:106886. doi: 10.1016/j.nedt.2025.106886. Epub 2025 Oct 5. PMID 41075434